CLINICAL TRIAL: NCT03659695
Title: Cardioprotective Effects of Freeze Dried Grape Powder Supplementation on Blood Pressure and Plasma Lipids/Lipoproteins: A Pilot Study
Brief Title: Cardioprotective Effects of Freeze Dried Grape Powder on Blood Pressure and Plasma Lipids/Lipoproteins
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Contract terminated
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Ann Skulas-Ray, Assistant Professor of Nutritional Sciences, University of Arizona
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Grape Study
Record Dates: First submitted 2018-09-02; First posted 2018-09-06 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Cardiovascular Risk Factor
MeSH Terms: interventions — whole grape extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grape Powder (Experimental): 69 g/d freeze dried grape powder
  Interventions: Dietary Supplement: Grape Powder
- Placebo powder (Placebo Comparator): 69 g/d placebo powder matched for taste and appearance
  Interventions: Dietary Supplement: Placebo Powder

INTERVENTIONS:
Dietary Supplement: Grape Powder — 69 g/d freeze dried grape powder
  Arms: Grape Powder
Dietary Supplement: Placebo Powder — 69 g/d placebo powder matched for taste and appearance
  Arms: Placebo powder

SUMMARY:
Whole food-based dietary interventions have the potential to promote cardiometabolic health via multiple mechanisms, including improvements in blood pressure, bad cholesterol, and other markers of metabolic health. Previous research suggests that grapes have the potential to promote optimal cardiometabolic function by reducing LDL-C, but it remains unclear whether there is a dose-response relationship. Moreover, few studies have evaluated effects on vascular health following daily grape consumption. We propose to examine the effects of 6-8 weeks of supplementation with freeze dried grape powder (69 g/d; ~three ¾ cup servings) compared to a control powder without grapes on: 1) bad cholesterol and blood pressure and 2) other measures of cardiometabolic health, including glucose and insulin. We will enroll overweight (BMI 25-36 kg/m2) but otherwise healthy adults with moderately elevated LDL-C (>115 mg/dL for women and >130 mg/dL for men) and/or blood pressure of120-159/80-99 mm Hg. This will optimize the potential for observing significant changes in these measures of health. We will recruit 20 eligible participants with the expectation that at least 15 will complete the study. The placebo-controlled, crossover study design will allow for a direct comparison of effects within the same participant. We anticipate that the bioactive components of grapes will promote cardiometabolic health via changes in LDL-C and blood pressure. Results from the proposed study would help to clarify how daily grape consumption might promote health and would provide further support for incorporating whole, unprocessed fruit in a healthy dietary pattern.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 25-36 kg/m2
* At least one of the following:

  * LDL-C above 115 mg/dL (women) or above 130 mg/dL (men)
  * Systolic blood pressure of 120-159 mmHg
  * Diastolic blood pressure of 80-99 mmHg

Exclusion Criteria:

* Allergies to grapes
* History of CVD, blood pressure ≥ 160/100 mmHg, kidney disease, diabetes, or inflammatory diseases such as GI disorders and rheumatoid arthritis
* Use of medications/supplements for elevated lipids, blood pressure, or glucose
* Chronic use of non-steroidal anti-inflammatory or immunosuppressant drugs
* Conditions requiring chronic use of steroids

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2024-02-13 (Actual)

PRIMARY OUTCOMES:
LDL-C/non-HDL-C | 6-8 weeks
Brachial and central blood pressure | 6-8 weeks
  systolic and diastolic pressures

SECONDARY OUTCOMES:
Pulse Wave Velocity (PWV) | 6-8 weeks
Augmentation Index | 6-8 weeks
  augmentation index corrected for heart rate
Other lipids and lipoproteins | 6-8 weeks
  HDL-C, total cholesterol, and triglycerides
Glucose | 6-8 weeks
  fasting blood glucose
Insulin | 6-8 weeks
  fasting blood insulin

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arizona Agricultural Center, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] U.S. Department of Health and Human Services and U.S. Department of Agriculture, 2015-2020 Dietary Guidelines for Americans, 2015.
- [Background] Zern TL, Wood RJ, Greene C, West KL, Liu Y, Aggarwal D, Shachter NS, Fernandez ML. Grape polyphenols exert a cardioprotective effect in pre- and postmenopausal women by lowering plasma lipids and reducing oxidative stress. J Nutr. 2005 Aug;135(8):1911-7. doi: 10.1093/jn/135.8.1911. PMID 16046716
- [Background] Seymour EM, Singer AA, Bennink MR, Parikh RV, Kirakosyan A, Kaufman PB, Bolling SF. Chronic intake of a phytochemical-enriched diet reduces cardiac fibrosis and diastolic dysfunction caused by prolonged salt-sensitive hypertension. J Gerontol A Biol Sci Med Sci. 2008 Oct;63(10):1034-42. doi: 10.1093/gerona/63.10.1034. PMID 18948553
- [Background] Patki G, Allam FH, Atrooz F, Dao AT, Solanki N, Chugh G, Asghar M, Jafri F, Bohat R, Alkadhi KA, Salim S. Grape powder intake prevents ovariectomy-induced anxiety-like behavior, memory impairment and high blood pressure in female Wistar rats. PLoS One. 2013 Sep 9;8(9):e74522. doi: 10.1371/journal.pone.0074522. eCollection 2013. PMID 24040270
- [Background] Allam F, Dao AT, Chugh G, Bohat R, Jafri F, Patki G, Mowrey C, Asghar M, Alkadhi KA, Salim S. Grape powder supplementation prevents oxidative stress-induced anxiety-like behavior, memory impairment, and high blood pressure in rats. J Nutr. 2013 Jun;143(6):835-42. doi: 10.3945/jn.113.174649. Epub 2013 Apr 17. PMID 23596160
- [Background] Thandapilly SJ, LeMaistre JL, Louis XL, Anderson CM, Netticadan T, Anderson HD. Vascular and cardiac effects of grape powder in the spontaneously hypertensive rat. Am J Hypertens. 2012 Oct;25(10):1070-6. doi: 10.1038/ajh.2012.98. Epub 2012 Jul 12. PMID 22785408
- [Background] Perez-Jimenez J, Saura-Calixto F. Grape products and cardiovascular disease risk factors. Nutr Res Rev. 2008 Dec;21(2):158-73. doi: 10.1017/S0954422408125124. PMID 19087369
- [Background] Rasines-Perea Z, Teissedre PL. Grape Polyphenols' Effects in Human Cardiovascular Diseases and Diabetes. Molecules. 2017 Jan 1;22(1):68. doi: 10.3390/molecules22010068. PMID 28045444
- [Background] Chaves AA, Joshi MS, Coyle CM, Brady JE, Dech SJ, Schanbacher BL, Baliga R, Basuray A, Bauer JA. Vasoprotective endothelial effects of a standardized grape product in humans. Vascul Pharmacol. 2009 Jan-Feb;50(1-2):20-6. doi: 10.1016/j.vph.2008.08.004. Epub 2008 Sep 7. PMID 18805507
- [Background] Barona J, Aristizabal JC, Blesso CN, Volek JS, Fernandez ML. Grape polyphenols reduce blood pressure and increase flow-mediated vasodilation in men with metabolic syndrome. J Nutr. 2012 Sep;142(9):1626-32. doi: 10.3945/jn.112.162743. Epub 2012 Jul 18. PMID 22810991
- [Background] Zunino SJ, Peerson JM, Freytag TL, Breksa AP, Bonnel EL, Woodhouse LR, Storms DH. Dietary grape powder increases IL-1beta and IL-6 production by lipopolysaccharide-activated monocytes and reduces plasma concentrations of large LDL and large LDL-cholesterol particles in obese humans. Br J Nutr. 2014 Aug 14;112(3):369-80. doi: 10.1017/S0007114514000890. Epub 2014 May 15. PMID 24832727
- [Background] Ridker PM, Rifai N, Cook NR, Bradwin G, Buring JE. Non-HDL cholesterol, apolipoproteins A-I and B100, standard lipid measures, lipid ratios, and CRP as risk factors for cardiovascular disease in women. JAMA. 2005 Jul 20;294(3):326-33. doi: 10.1001/jama.294.3.326. PMID 16030277
- [Background] Jacobson TA, Maki KC, Orringer CE, Jones PH, Kris-Etherton P, Sikand G, La Forge R, Daniels SR, Wilson DP, Morris PB, Wild RA, Grundy SM, Daviglus M, Ferdinand KC, Vijayaraghavan K, Deedwania PC, Aberg JA, Liao KP, McKenney JM, Ross JL, Braun LT, Ito MK, Bays HE, Brown WV, Underberg JA; NLA Expert Panel. National Lipid Association Recommendations for Patient-Centered Management of Dyslipidemia: Part 2. J Clin Lipidol. 2015 Nov-Dec;9(6 Suppl):S1-122.e1. doi: 10.1016/j.jacl.2015.09.002. Epub 2015 Sep 18. PMID 26699442
- [Background] McEniery CM, Cockcroft JR, Roman MJ, Franklin SS, Wilkinson IB. Central blood pressure: current evidence and clinical importance. Eur Heart J. 2014 Jul;35(26):1719-25. doi: 10.1093/eurheartj/eht565. Epub 2014 Jan 23. PMID 24459197
- [Background] Ben-Shlomo Y, Spears M, Boustred C, May M, Anderson SG, Benjamin EJ, Boutouyrie P, Cameron J, Chen CH, Cruickshank JK, Hwang SJ, Lakatta EG, Laurent S, Maldonado J, Mitchell GF, Najjar SS, Newman AB, Ohishi M, Pannier B, Pereira T, Vasan RS, Shokawa T, Sutton-Tyrell K, Verbeke F, Wang KL, Webb DJ, Willum Hansen T, Zoungas S, McEniery CM, Cockcroft JR, Wilkinson IB. Aortic pulse wave velocity improves cardiovascular event prediction: an individual participant meta-analysis of prospective observational data from 17,635 subjects. J Am Coll Cardiol. 2014 Feb 25;63(7):636-646. doi: 10.1016/j.jacc.2013.09.063. Epub 2013 Nov 13. PMID 24239664
- [Background] Woerdeman J, van Poelgeest E, Ket JCF, Eringa EC, Serne EH, Smulders YM. Do grape polyphenols improve metabolic syndrome components? A systematic review. Eur J Clin Nutr. 2017 Dec;71(12):1381-1392. doi: 10.1038/ejcn.2016.227. Epub 2017 Feb 1. PMID 28145414